CLINICAL TRIAL: NCT04864015
Title: COVID-19: a Study About Aerosol Formation During Gastroscopy With a Adjusted Mouthpiece for Droplet Reduction
Brief Title: COVID-19 Aerosol in EGD Using a Droplet Reduction Mouthpiece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: s65197
Record Dates: First submitted 2021-04-27; First posted 2021-04-28 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Droplet Spread; Covid19
Keywords: droplet reduction mask; COVID-19; upper GI endoscopy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A investigator-initiated single center open-label randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional mouthpiece (Placebo Comparator): Patients undergoing standard EGD using a conventional mouthpiece
  Interventions: Device: Mouthpiece B1(Mouthpiece MPC-ST GMDN:62534 Generic name: Endoscopic bite block, basic, reusable
- Droplet reduction mouthpiece (Active Comparator): Patients undergoing standard EGD using a new droplet reduction mouthpiece
  Interventions: Device: Mouthpiece B1(Mouthpiece MPC-ST GMDN:62534 Generic name: Endoscopic bite block, basic, reusable

INTERVENTIONS:
Device: Mouthpiece B1(Mouthpiece MPC-ST GMDN:62534 Generic name: Endoscopic bite block, basic, reusable — Use of a Mouthpiece B1 during standard EGD instead of a conventional mouthpiece

SUMMARY:
Measurement of aerosolisation during esophagogastroduodenoscopy (EGD) to compare two types of mouthpieces, conventional versus a new and commercially available one 'the droplet reduction mouthpiece B1'.

This new mouthpiece is considered to reduce droplet spreading during EGD and therefore could be a good option for use in COVID-19 positive patients.

DETAILED DESCRIPTION:
During esophagogastroduodenoscopy (EGD), a hard-plastic mouthpiece is used to protect the endoscope from being bitten and to enable its smooth insertion. In September 2020, the droplet reduction Mouthpiece "B1" (Mouthpiece MPC-ST GMDN:62534 Generic name: Endoscopic bite block, basic, reusable) was launched by Fujifilm Corporation, Tokyo, Japan and imported to Europe by Fujifilm Europe. The droplet reduction mouthpiece is used in the same way as the conventional mouthpiece but differs from current mouthpieces by the inclusion of a sponge rubber incorporated into the mouthpiece orifice, and a drape shield specifically created to catch and reduce the droplets emitted by the patient during upper gastrointestinal endoscopy. This newly developed mouthpiece is considered for application during routine endoscopy at our facility during the COVID-19 pandemic, helping to minimize the risk to health care workers and patients from becoming infected with COVID-19 and various other pathogens. However, there is a lack of scientific evidence on the amount of aerosol reduction with the modified mouthpiece when upper gastrointestinal (GI) endoscopy is being performed.

The aim of the present study is to quantify the generation of aerosols when performing upper GI endoscopy with the modified mouthpiece. The investigators intend to quantify the number of particles in the air near the patient. The duration of therapeutic upper gastrointestinal endoscopies can vary extremely. To avoid risk of imbalance in procedure durations, the investigational team is limiting the protocol to standard diagnostic EGDs. The investigators assume that aerosol generations during short procedures can be extrapolated to longer procedures and hence this should not invalidate the findings

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old;
* Male or female patients;
* Patients undergoing elective standard diagnostic EGD;
* Negative polymerase chain reaction (PCR) test on nasopharyngeal swab 24 or 48 hours prior to the test;
* No anatomical deformity of nose and throat, no known diseases of nose and throat;
* Signed informed consent

Exclusion Criteria:

* Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Generation of aerosol particles by esophagogastroduodenoscopy with the droplet reduction mouthpiece. | 4 months
  Number of aerosols generated by EGD with the droplet reduction mouthpiece

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — UZ Leuven, KU Leuven; Raf Bisschops, MD, PhD, Principal Investigator — UZ Leuven, KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
We won't share individual participant data

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT04864015/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT04864015/ICF_001.pdf